CLINICAL TRIAL: NCT05667467
Title: Investigation of the Effect of Care Bundle Implementation on Recovery Process in Open Heart Surgery Patients
Brief Title: The Effect of Care Bundle in Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Yasemin Yılmaz, Lecturer, Harran University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: Harran University
Record Dates: First submitted 2022-12-07; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Thoracic Surgery; Patient Care Bundles
Keywords: Patient care bundles; Nursing; Perioperative nursing; Cardiac surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL GROUP (Experimental)
  Interventions: Procedure: Care Bundle Implementation
- NURSE GROUP (Experimental)
  Interventions: Procedure: Care Bundle Implementation
- STUDY GROUP (Experimental)
  Interventions: Procedure: Care Bundle Implementation

INTERVENTIONS:
Procedure: Care Bundle Implementation — In this study, the control group received standard care. The nurse group was given training on the implementation of the care bundle. A "cardiac surgery care bundle" was applied to the study group by clinical nurses.

SUMMARY:
This study is a quasi-experimental (non-randomized) design study with control and study group patients undergoing open heart surgery. The main purpose of the research to examine the effect of the care bundle application on the quality of recovery and respiratory patterns (respiratory rate, presence of dyspnea, oxygen saturation, etc.) in patients with open heart surgery. The other purpose is examine the compliance rates of nurses in the implementation of the cardiac surgery care bundle on patients. In the study, nurses working in the cardiovascular surgery clinic and surgical intensive care unit in a training and research hospital in southeast Turkey voluntarily applied the care bundle created by the researcher to the patients in the study group. When the data of the study were examined, it was seen that the respiratory patterns and recovery status of the patients who received the care bundle were better. However, it was determined that the compliance rate of the nurses to the care bundle was not at the desired level.

DETAILED DESCRIPTION:
Introduction: There are several ways to transfer evidence-based practice to the clinic. One of them is "care bundle" implementation.

Purpose: To examine the effect of applying the "Cardiac Surgery Care Bundle" which consists of evidence-based applications, on patients with open heart surgery (AKC) on the quality of recovery and respiratory patterns (respiratory rate, presence of dyspnea, oxygen saturation, etc.). In the study, the compliance status of nurses in the implementation of the care bundle was also examined.

Method:This research is a quasi-experimental, non-randomized study with AKC applied control and study groups. In the study, volunteer nurses working in the surgical intensive care and cardiovascular surgery clinics applied the care bundle created by the researcher to the patients in the study group. care bundle; It includes "Informing the Patients and Their Relatives", "Respiratory Management" and "Early Mobilization" implementations. A total of 103 patients, 69 of whom were control and 34 were study, were included in the study. First, the data of the control group and then the study group were collected. Patients in the control group received standard care, while the study group received a care bundle in addition to the standard care. Data were obtained using the "Descriptive Characteristics Data Form", "Patient Outcomes for Complications Form" and the "Quality of Recovery-40-QoR-40".

Statistical analyses were performed using the IBM SPSS for Windows 22.0 software. The variables were analyzed for normality of distribution using skewness and kurtosis coefficients. Normally distributed variables were presented using mean ± standard deviation values and non-normally distributed variables were presented using median (minimum-maximum) values. Differences between two samples were analyzed using the "Independent Samples t test" when the assumption of normality was met, and using the "Mann-Whitney U" test when the assumption of normality was not met. Categorical variables were analyzed using Chi-square or Fisher's exact tests. Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Patients

  * 18 years and older,
  * Elective AKC planned
  * Those who will undergo cardiac surgery for the first time
  * Extubated after cardiac surgery and not given sedating drugs
  * No communication barrier (including hearing and vision problems),
  * Does not have a musculoskeletal disease or neurological problem that will prevent walking after surgery,
  * Does not have any respiratory disease,
  * Psychiatric, not diagnosed with mental illness,
  * Those who volunteered to participate in the research
  * Patients who are 18 years of age or older who volunteer to participate in the research.
* Inclusion Criteria for Nurses

  * Working as a nurse in cardiovascular surgery clinic or surgical intensive care clinic,
  * It is the nurses who volunteer to participate in the research.

Exclusion Criteria:

* Exclusion Criteria for Patients

  * Patients with active bleeding after surgery
  * Developing neurological complications
  * Complications that prevent the patient from standing up after surgery
  * Those with respiratory problems that will delay weaning from the mechanical ventilator
  * Re-operated due to the development of any complication
  * Those who want to leave the research during the pre- or post-surgical research process
  * These are the patients who develop a situation where they cannot continue to accompany the patient while they are accompanying the patient, or who are the relatives of the patients who want to leave the research during the research process.
* Exclusion Criteria for Nurses

  * Assigned to another clinic during the research process,
  * Resigned from his job during the research process,
  * Nurses who want to leave the study during any phase of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
The effect of the care bundle on the recovery status of the patients | One week after surgery
  In the study, the recovery status of patients after surgery was measured with the "Recovery Quality-40 Questionnaire". The contribution of the cardiac surgery care bundle applied to the study group by the clinical nurses to the recovery status was examined.

SECONDARY OUTCOMES:
Examination of nurses' compliance with the care bundle | One week after the data collection process of the study group patients was completed.
  In this study, nurses' compliance rates to the care bundle (application rates to patients) were examined. According to the literature, compliance should be at least 95% in order to have a high level of compliance with the care bundle.

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin Yılmaz, Sanliurfa, Haliliye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Moradian ST, Najafloo M, Mahmoudi H, Ghiasi MS. Early mobilization reduces the atelectasis and pleural effusion in patients undergoing coronary artery bypass graft surgery: A randomized clinical trial. J Vasc Nurs. 2017 Sep;35(3):141-145. doi: 10.1016/j.jvn.2017.02.001. PMID 28838589
- [Background] Zanini M, Nery RM, de Lima JB, Buhler RP, da Silveira AD, Stein R. Effects of Different Rehabilitation Protocols in Inpatient Cardiac Rehabilitation After Coronary Artery Bypass Graft Surgery: A RANDOMIZED CLINICAL TRIAL. J Cardiopulm Rehabil Prev. 2019 Nov;39(6):E19-E25. doi: 10.1097/HCR.0000000000000431. PMID 31343586
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Buerge M, Magboo R, Wills D, Karpouzis I, Balmforth D, Cooper P, Roberts N, O'Brien B. Doing Simple Things Well: Practice Advisory Implementation Reduces Atrial Fibrillation After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2913-2920. doi: 10.1053/j.jvca.2020.06.078. Epub 2020 Jul 3. PMID 32741608
- [Background] Meersch M, Schmidt C, Hoffmeier A, Van Aken H, Wempe C, Gerss J, Zarbock A. Prevention of cardiac surgery-associated AKI by implementing the KDIGO guidelines in high risk patients identified by biomarkers: the PrevAKI randomized controlled trial. Intensive Care Med. 2017 Nov;43(11):1551-1561. doi: 10.1007/s00134-016-4670-3. Epub 2017 Jan 21. PMID 28110412